CLINICAL TRIAL: NCT01430221
Title: Mindfulness-based Personalized Health Planning for Reducing Risk of Heart Disease and Diabetes
Acronym: AWARENESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00016540; R01HL067459 (NIH)
Record Dates: First submitted 2011-09-02; First posted 2011-09-08 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Prediabetes; Depressive Symptoms Mild to Moderate in Severity
Keywords: prediabetes; severity of depressive symptoms; mindfulness; personalized health planning; cardiometabolic diseases prevention
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MB-PHP Group (Experimental): Mindfulness-based Personalized Health Planning (MB-PHP)with health coaching. MB-PHP includes weekly small group meetings for 22-weeks and 10 bi-weekly telephonic health coaching.
  Interventions: Behavioral: Mindfulness-based Personalized Health Planning
- SAGE Group (Active Comparator): Structure & Guided Education (SAGE) includes small group-education sessions once per week for 22 weeks. Subjects also participate in 10 bi-weekly telephone calls with education partners who use supportive listening techniques..
  Interventions: Other: Structured & Guided Education

INTERVENTIONS:
Behavioral: Mindfulness-based Personalized Health Planning
  Other Names: MB-PHP
  Arms: MB-PHP Group
Other: Structured & Guided Education
  Other Names: SAGE
  Arms: SAGE Group

SUMMARY:
The purpose of this study is to compare the effectiveness of educational and lifestyle intervention programs aimed at reducing fasting blood sugar and emotional distress in adults with prediabetes.

DETAILED DESCRIPTION:
There is a need for the development of new preventive strategies to help combat the rising prevalence of type 2 diabetes (T2D) and coronary heart disease (CHD). This need is particularly critical for individuals who already show impaired fasting glucose (IFG) which incurs a greater risk of T2D and CHD than those with normal glucose levels. Lifestyle changes are effective in reducing fasting glucose although changes in behaviors are challenging and may be more so among individuals with symptoms of depression. Evidence suggests that elevated symptoms of depression significantly impacts adiposity, levels of inflammatory biomarkers, and other early risk factors of cardiometabolic conditions. With few exceptions, current lifestyle interventions are 'one-size fits all' and pay little or no attention to patients' individual goals, resources, and barriers to making positive behavior changes with no lifestyle intervention addressing patients current mental states. By adopting a 'patient-centered' strategy, this study will test the effectiveness of a Mindfulness-based Personalized health planning (MB-PHP) in persons with prediabetes (e.g., defined by hemoglobin (h) A1c of 5.7%-6.4% and elevated symptoms of depression. The MB-PHP incorporates four primary strategies: (1) individual risk quantification of T2D and cardiovascular disease (CVD) based on hA1c and level of depressive symptoms; (2) group-based education on behavioral and traditional risk factors for CVD and T2D; (3) development of a personalized health plan (PHP) that emphasizes lifestyle areas where the patient is willing and ready to change; and (4) support in PHP implementation and patient engagement through integrative health partnering. To further support the goals of the PHP, mindfulness meditation is used to promote greater awareness of the unity of mind and body and specifically how unconscious thoughts, feelings, and behaviors can undermine achieving healthy lifestyle behaviors. The MB-PHP emphasizes personalize, predictive, and preventive risk management while fostering meaningful subject engagement with the goal of reducing fasting glucose and depressive symptom severity.

ELIGIBILITY:
Inclusion Criteria:

1. Between 30 and 70 years old 2. Nonsmoker 3. Generally in good health 4. Able to speak and read English 5. Willing to provide informed consent 6. Patient Health Questionnaire-9 (PHQ-9) score greater than 5 (minimal depression) but less than 25 (severe depression) 7. Hemoglobin A1c values between 5.6%-6.4% (inclusive) 9. Able to attend 2 study visits at Duke University Medical Center 10. Able to attend 22 small group education sessions 11. Able to participate in 10 telephonic support sessions

Exclusion Criteria:

1. Younger than 30 years old/Older than 70
2. PHQ-9 score of 25 or greater (severe depression) and lower than 5 (no depression)

4. Hemoglobin A1c below 5.6% or above 6.4% 5. BMI less than 19.1 kg/m2 6. History of cardiovascular diseases (e.g., coronary artery disease, congestive heart failure, prior myocardial infarction or stroke, or more than 4 episodes of chest pain requiring nitroglycerin in the last month) 7. Current smokers or former smokers who quit within the last 6 months 8. Participation in formal group exercise, nutrition, weight loss or stress management program during the study period 9. Severe disease that may make cardiovascular prevention of secondary importance and/or result in severely compromised immune system (e.g., HIV positive, end-stage renal disease requiring dialysis, Hepatitis C) 10. Terminal illness defined as requiring oxygen or diagnosis of malignancy 11. Unstable medical conditions underlying weight or eating problems (e.g., Cushing's Syndrome, thyroid disorder) 12. Use of medications that impact immune, cardiovascular, or metabolic indices (e.g., anti-inflammatory, anti-hypertensives, lipid-lowering medications, oral agents for diabetes, stimulants) 13. Women on exogenous hormone replacement or oral contraceptives 14. Women reporting irregular menstrual cycle over previous 6 months 15. Severe psychiatric conditions or behaviors (e.g., drug or alcohol abuse, psychosis, severe social anxiety, bipolar disorder, Axis II diagnosis) 16. Unwillingness to accept randomization 17. Pregnancy

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2011-05; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Fasting glucose | screening, up to 45-days after completion of intervention, long term follow-up (>6 months)
  Changes from entry levels of fasting glucose up to 45-days post-intervention, and long-term follow-up (>6-months) levels.
Severity of depressive symptoms | baseline, up to 45-days after completion of intervention, long-term follow-up (>6 months)
  Changes from entry levels of severity of depressive symptoms as assessed via the Hamilton Depression (HAM-D) interview to 45-days after completion of intervention and long-term follow-up (> 6-months)

SECONDARY OUTCOMES:
Reduction in resting blood pressure | Baseline, up to 45-days after completion of intervention, long-term follow-up (>6 months)
  Changes in systolic and diastolic blood pressure 45-days following completion of intervention and long-term follow-up.
Changes in inflammation | baseline, 45-days following completion of intervention and long-term follow-up(>6-months)
  Pre-to-post changes in inflammation as assessed by high sensitivity C-reactive protein (hsCRP) and in vitro production of stimulated cytokines 45-days following completion of intervention and long-term follow-up..

CONTACTS AND LOCATIONS:
Overall Officials: Edward Suarez, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States